CLINICAL TRIAL: NCT01095744
Title: Influence of Age on amyloïd Load in Alzheimer's Disease and in Atypical Focal Cortical Alzheimer's Disease Like Posterior Cortical Atrophy (PCA) and Logopenic Progressive Aphasia (LPA)Using Positron Emitting Tomography (PET) Imaging
Brief Title: Influence of Age on Amyloid Load in Alzheimer's Disease and in Atypical Focal Cortical Alzheimer's Disease
Acronym: BIOMAGE
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C08-30; 2008-A00939-46 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-03-12; First posted 2010-03-30 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2012-02

CONDITIONS: Alzheimer's Disease; Posterior Cortical Atrophy; Logopenic Progressive Aphasia
Keywords: PIB imaging,; brain atrophy; cognitive impairment; Pet imaging; Alzheimer's disease; amyloid protein
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Amyloidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA sample immortalized blood cell cultures csf aliquots for patients who beneficiated from a lumbar puncture.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- EOAD typical AD: this cohort is constituted with early onset typical AD.
- LOAD typical: this group is constituted with late onset typical AD
- atypical AD: this group is constituted with atypical form of focal cortical atrophy, like posterior cortical atrophy and logopenic progressive aphasia.
- young controls: under 65
- old controls: over 65

SUMMARY:
The first objective is to asses influence of age on amyloid load measured by PET imaging using Pittsburgh B compound (PiB) radio-tracer, in Alzheimer's disease(AD). This will allow the determination of brains age-specific deterioration factors by comparing Early onset AD (EOAD), Late onset AD (LOAD)and atypical focal cortical AD (PCA and LPA). The amount of brain lesions in AD patients is estimated by:

1. measuring the rate of cortical brain atrophy,
2. FDG imaging of glucose metabolism reflecting neuronal activity, and
3. for patients who benefited from a lumbar puncture; Cortical-spinal fluid (CSF) amounts of amyloïd and tau proteins are measured.

DETAILED DESCRIPTION:
Literature data suggests there are different types of AD depending on their age of onset, called EOAD and LOAD. These two categories are distinguished by the localization of brain atrophy : severe and 'posterior' in EOAD and more 'anterior' in LOAD. Neuro-pathologic data suggests some atypical focal cortical atrophy, characterized by a respect of episodic memory, may be classified within EOAD.

PiB-based PET imaging allows the in-vivo visualization and quantification of amyloïd load.

We want to answer the question whether the amount of amyloïd protein may be lower in LOAD than EOAD in patients showing the same level of dementia, and thus identify ageing-specific cognitive disorders and understand witch factors influence etio-pathology of typical and atypical Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* AD patients: clinical dementia rating between 0.5 and 2 free and cued recall test (Grober and Buschke) cued-recall < 18/48 and total recall < 40/48
* atypical AD : i visual-spatial disorder and respect of episodic memory progressive evolution, Balint syndrome ii progressive language disorder constituted of logopenic aphasia respect of episodic memory
* controls: age over 30 MMSE over or equal to 27 normal neuropsychiatric state for age and education level

Exclusion Criteria:

* for every patients : psychiatric disorders age under18 absence of social security counter indication to MRI supposed or actual alcoholism or drug addiction pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients have to fulfil criteria for (1)AD with an amnesic syndrome of the media-temporal type, EOAD have lower frequency and (2) and for atypical Ad respecting episodic memory, inaugural language disorder or visual-spatial disorder
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
PIB-PET imaging of amyloid load | 0 - 2 months
  PET imaging using PIB radio-tracer will give an estimation of regional amyloid load for every patient
FDG-PET imaging of glucose metabolism | 0 - 2 months
  PET imaging using 18F-fluorodesoxyglucose (FDG) will give a visualization of regional neuronal metabolism
clinical phenotypic assessment | 0 - 2 months
  the clinical evaluation includes a neurologic consulting, a neuropsychologic assessment of cognitive performances, and evaluation of autonomy
MRI | 0 - 2 months
  the magnetic resonance imaging will be performed using numerous modalities like T1 weighted sequences for anatomic information, T2 weighted FLAIR and TSE sequences to avoid vascular injuries and T2 GRE to avoid microbleeds, DTI for the diffusion tensor imaging and default mode FMRI, to identify neural networks involved in default concious mode.
ApoE gene sequencing | 0 - 24 months after inclusion
  ApoE gene sequencing, will be performed after all samples have been collected. So this may be 0 to 24 month after inclusion.

SECONDARY OUTCOMES:
amyloid and Tau measurements in cerebro-spinal fluid (csf) | -6 months or +6months arround T0
  some patients have a lumbar puncture that allows a direct quantification of CSF amyloid, tau and phospho-tau amounts.This measure is performed in the 6 months following the clinical assessment (at inclusion) and when a former puncture has already been done, it can be used retro-actively up to 6 months before clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Dubois, professor doctor, Principal Investigator — INSERM U975; marie c sarzin, doctor, Study Chair — Inserm U975
Locations (1):
- Pitie Salpêtrière Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Dorothee G, Bottlaender M, Moukari E, de Souza LC, Maroy R, Corlier F, Colliot O, Chupin M, Lamari F, Lehericy S, Dubois B, Sarazin M, Aucouturier P. Distinct patterns of antiamyloid-beta antibodies in typical and atypical Alzheimer disease. Arch Neurol. 2012 Sep;69(9):1181-5. doi: 10.1001/archneurol.2012.604. PMID 22710357
- [Result] Migliaccio R, Agosta F, Toba MN, Samri D, Corlier F, de Souza LC, Chupin M, Sharman M, Gorno-Tempini ML, Dubois B, Filippi M, Bartolomeo P. Brain networks in posterior cortical atrophy: a single case tractography study and literature review. Cortex. 2012 Nov-Dec;48(10):1298-309. doi: 10.1016/j.cortex.2011.10.002. Epub 2011 Oct 20. PMID 22099855
- [Result] de Souza LC, Corlier F, Habert MO, Uspenskaya O, Maroy R, Lamari F, Chupin M, Lehericy S, Colliot O, Hahn-Barma V, Samri D, Dubois B, Bottlaender M, Sarazin M. Similar amyloid-beta burden in posterior cortical atrophy and Alzheimer's disease. Brain. 2011 Jul;134(Pt 7):2036-43. doi: 10.1093/brain/awr130. PMID 21705422